CLINICAL TRIAL: NCT03960879
Title: DNA Methylation Testing for the Screening of Uterine Cervical Lesion: A Prospective Cohort Study
Brief Title: DNA Methylation for Screening Uterine Cervical Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: METHY2
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: DNA Methylation; Uterine Cervical Cancer; High Grade Squamous Intraepithelial Lesions; Low Grade Squamous Intraepithelial Lesions
MeSH Terms: conditions — Uterine Cervical Neoplasms; Squamous Intraepithelial Lesions | interventions — DNA Methylation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Uterine cervical cytology collected during the clinical settings for the testing of DNA methylation, TCT and high-risk HPV
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DNA methylation — DNA methylation for the cervical cytology
Diagnostic Test: High-risk HPV — High-risk HPV testing for the cervical cytology
Diagnostic Test: TCT — Thin prep liquid-based cytology test for the cervical cytology

SUMMARY:
The primary objective of this study is to compare the testing of DNA methylation, high-risk HPV subtypes, and cytology with the definite histological results for uterine cervical lesions in a prospective cohort study.

This study will include 300 unselected patients with definite histological results. All the cervical specimens of cytology collected in the clinical settings will be utilized for the testing of DNA methylation, high-risk HPV subtypes and thin prep liquid-based cytology test (TCT). The sensitivity, specificity, positive predictive value and negative predictive value were calculated based on the known histological results. The differences of DNA methylation with high-risk human papillomavirus (HPV) and TCT will also be analyzed.

The testing of DNA methylation will be performed with the methylation-specific polymerase chain reaction (PCR). The TCT and HPV testing will be performed with the Roche kits.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cervical histology within one month when collecting cervical cytology
* Aged 18 years or older
* Signed an approved informed consents

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Confirmed cervical histology within one month when collecting cervical cytology
  * Aged 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of DNA methylation | 1 year
  Sensitivity of DNA methylation compared with histological results for the differentiation of cervical cancer and high grade squamous intraepithelial lesions (HSIL)
Specificity of DNA methylation | 1 year
  Specificity of DNA methylation compared with histological results for the differentiation of cervical cancer and HSIL

SECONDARY OUTCOMES:
Positive predictive value of DNA methylation | 1 year
  Positive predictive value of DNA methylation compared with histological results for the differentiation of cervical cancer and HSIL
Negative predictive value of DNA methylation | 1 year
  Negative predictive value of DNA methylation compared with histological results for the differentiation of cervical cancer and HSIL
Correlation coefficient of DNA methylation with other screening methods | 1 year
  Correlation coefficient of DNA methylation with high-risk HPV and TCT results

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided